CLINICAL TRIAL: NCT06541977
Title: The Effects of a Physical Activity Program Before and After Bariatric Surgery for People With Obesity: Referral From Healthcare Settings to the B-FIT Programme.
Brief Title: A New Model of Exercise Referral Scheme Before and After Bariatric Surgery for People With Obesity
Acronym: B-FIT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fundació Universitària del Bages (Other)
Collaborators: Althaia Xarxa Assistencial Universitària de Manresa (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: UManresa_B-FIT2024
Record Dates: First submitted 2024-07-30; First posted 2024-08-07 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: Obesity; Quality of Life; Weight Loss
Keywords: bariatric surgery; physical activity; quality of life; obesity
MeSH Terms: conditions — Obesity; Weight Loss; Motor Activity | interventions — Exercise; Bariatric Surgery

STUDY DESIGN:
Intervention Model Description: Groups will be followed and assessed concurrently but separately, ensuring that the comparison between interventions is clear and not influenced by crossover effects.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Pre and Post Intervention (Experimental): Participants in this group will receive the usual hospital care, which includes psychology visits, nutritional advice, and a physical activity protocol plan. In addition, participants will be referral form the Hospital to the Unviersity to undertake supervised physical activity sessions and health behavior change techniques aimed at reducing sedentary behavior and improving quality of life. This intervention will start 8 months before surgery and continue for 12 months post-surgery, with regular monitoring and support to sustain life-changing behaviors.
  Interventions: Behavioral: Behavioral to reduce sedentary behvaior; Behavioral: Physical activity; Procedure: Bariatric Surgery
- Post Intervention (Experimental): Participants in this group will receive the usual hospital care, including psychology visits, nutritional advice, and a physical activity protocol plan. Additionally, participants in this group will be referral from the Hospital to the Unviersity to begin supervised physical activity sessions and health behavior change techniques 12 months post-surgery, designed to reduce sedentary behavior and improve quality of life, with continuous professional support throughout the intervention period.
  Interventions: Behavioral: Behavioral to reduce sedentary behvaior; Behavioral: Physical activity; Procedure: Bariatric Surgery
- Comparision (Active Comparator): Participants in this group will receive the usual hospital care, which includes psychology visits, nutritional advice, and a physical activity protocol plan provided on a sheet. There will be no additional supervised physical activity sessions or health behavior change techniques beyond the standard care currently provided by the hospital.
  Interventions: Procedure: Bariatric Surgery

INTERVENTIONS:
Behavioral: Behavioral to reduce sedentary behvaior — This intervention will also utilize a geographical time app to raise awareness about participants' sedentary lifestyles, helping them identify opportunities to incorporate more movement into their daily routines. Furthermore, the program will implement the Wheel of Change behavior technique, which serves as a structured approach to facilitate lasting changes in health behaviors, empowering participants to take control of their physical activity levels and overall well-being.
  Arms: Post Intervention; Pre and Post Intervention
Behavioral: Physical activity — This intervention will be conducted with two weekly days of supervised and structured physical activity sessions, held at the university's facilities, providing participants with expert guidance and a supportive environment to enhance their physical fitness and overall health.
  Arms: Post Intervention; Pre and Post Intervention
Procedure: Bariatric Surgery — In this intervention, bariatric surgery will be performed, accompanied by the usual hospital care, which includes comprehensive nutritional and physical activity advice. This standard care ensures that participants receive essential guidance and support for their dietary and exercise routines, complementing the surgical intervention.

SUMMARY:
Obesity, defined by the WHO as an abnormal or excessive accumulation of fat that presents a risk to health, has reached pandemic levels, affecting approximately one-third of the world's population. This increase spans all ages, sexes, and socioeconomic levels, though it is more prevalent in older individuals and women.

Obesity is caused by an imbalance between energy intake and expenditure, influenced by genetic, epigenetic, social, and environmental factors. Key drivers are changes in the global food system, increased sedentary behavior, and reduced physical activity.

Complications include type II diabetes, myocardial infarction, various cancers, immune system problems, and increased mortality. Obesity also results in significant economic costs, with healthcare expenses 32% higher than for people of normal weight.

Bariatric surgery is the most effective long-term treatment for severe obesity, helping reduce body weight significantly in the first years post-surgery and improving metabolic control. However, individuals often regain weight in the long term. Factors influencing this include genetics, gastrointestinal hormones, adherence to diet, and healthy behaviors like physical activity.

Sedentary behavior and physical activity are crucial for maintaining weight loss post-surgery. Physical activity increases weight loss by 4% and improves outcomes when performed before surgery. However, lack of professional support, accessibility to sports facilities, and low socioeconomic status make it difficult to sustain these behaviors with simple advice alone.

Despite this, hospital interventions often focus solely on diet, offering only advice on physical activity. Effective interventions require supervised programs of more than six months to achieve long-term behavior changes.

The B-FIT (Bariatric surgery and FITness) project aims to create a new referral and intervention model for physical activity and reducing sedentary behavior in people with obesity before and after bariatric surgery. This model seeks to prevent post-surgery weight regain and promote healthy

DETAILED DESCRIPTION:
Obesity, as defined by the World Health Organization (WHO) as an abnormal or excessive accumulation of fat that presents a risk to health, has reached pandemic levels. Since 1980, its prevalence has doubled, affecting approximately one-third of the world's population. This increase spans all ages and both sexes, regardless of geographic location, ethnic origin, or socioeconomic level, though it is more prevalent in older individuals and women.

Obesity is a complex multifactorial disease primarily caused by an imbalance between energy intake and expenditure. Genetic, epigenetic, social, and microenvironmental factors contribute to its development. The main drivers of this pandemic are changes in the global food system, increased sedentary behavior, and reduced physical activity.

Complications and comorbidities associated with obesity include nearly all non-communicable diseases, such as type II diabetes, myocardial infarction, various types of cancer, immune system problems, and increased mortality in adulthood. Obesity also poses a significant economic cost, with 32% higher healthcare expenses compared to people of normal weight, divided into 31.8% direct costs and 68.2% indirect costs.

Currently, the most effective and cost-efficient long-term treatment for weight loss in people with obesity and comorbidities, or severe obesity, is bariatric surgery. Bariatric surgery is cost-effective, especially in the long term, helping to reduce body weight in the first years after the intervention (56.7% for gastric bypass and 45.9% for gastric balloon in the first ten years), improving metabolic control, and reducing obesity-related comorbidities.

However, individuals undergoing gastric bypass or gastric balloon surgery tend to regain weight in the long term. At least one in six operated individuals regain weight, and by 24 months post-surgery, up to 50% of patients regain weight. Factors such as genetics, anatomy, gastrointestinal hormones, adherence to a balanced diet, and healthy behaviors (reducing sedentary behavior and increasing physical activity) influence weight regain after bariatric surgery.

Sedentary behavior and physical activity are crucial for maintaining weight loss post-bariatric surgery. Physical activity post-surgery increases weight loss by 4%, and when performed before the intervention, improves weight loss at 12 months follow-up. However, the predisposition to obesity and weight regain post-surgery is influenced by factors such as lack of professional support, accessibility to sports facilities, and low socioeconomic status, making it difficult to improve physical activity levels and reduce sedentary behavior with simple health advice.

Despite this knowledge, hospital interventions before and after bariatric surgery focus on improving diet and only offer advice on physical activity, never physical activity and health behavior change interventions. Although diet is crucial and these interventions are often sufficient, physical activity and reducing sedentary behavior require supervised interventions of more than six months to achieve long-term behavior changes.

For these reasons, it is important to study through randomized clinical trials, with long-term follow-up, the effects of physical activity and reducing sedentary behavior on weight control, metabolic outcomes, and the quality of life, both mental and physical, of people with obesity who are going to undergo or have undergone bariatric surgery.

The B-FIT (Bariatric surgery and FITness) project aims to create a new referral and intervention model, from Hospital Sant Joan de Déu (Fundación Althaia) to the University of Vic-Central University of Catalonia, for physical activity and reducing sedentary behavior in people with obesity, both before and after bariatric surgery. This model aims to prevent post-surgery weight regain and promote healthy habits through behavior change techniques and supervised physical activity.

ELIGIBILITY:
Inclusion Criteria:

* Age: Adults aged 18-65 years.
* BMI: Body Mass Index (BMI) ≥ 35 kg/m² with associated comorbidities (e.g., type II diabetes, hypertension) or BMI ≥ 40 kg/m² without comorbidities.
* Eligibility for Bariatric Surgery: Candidates must be approved for bariatric surgery by their healthcare provider.
* Consent: Willingness to participate in the study, including signing an informed consent form.
* Commitment: Ability to commit to the study protocol, including pre-surgery and post-surgery interventions and follow-up assessments.
* Stable Medication: Participants must be on a stable medication regimen for any existing conditions for at least three months prior to the study.

Exclusion Criteria:

* Previous Bariatric Surgery: Individuals who have undergone any form of bariatric surgery previously.
* Medical Conditions: Presence of medical conditions that contraindicate physical activity, such as severe cardiovascular disease, uncontrolled hypertension, or orthopedic conditions that limit mobility.
* Psychiatric Disorders: Severe psychiatric disorders or substance abuse issues that might impair the ability to comply with the study protocol.
* Pregnancy: Pregnant or planning to become pregnant during the study period. Participation in Other Studies: Currently participating in another clinical trial or weight loss program.
* Non-compliance Risk: Any other condition or factor that the investigators believe would prevent the participant from complying with the study protocol or that would put the participant at risk.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2025-09-09 (Estimated); Primary Completion 2026-05-02 (Estimated); Study Completion 2036-06-30 (Estimated)

PRIMARY OUTCOMES:
Physical activity levels | Once a year during ten years
  Levels of Moderate to vigorous physical activity, light physical activity using accelerometry
Sedentary behavior patterns | Once a year during ten years
  Number and time of Sedentary bouts and breaks using accelerometry
Mass Body Index | Once a year during ten years
  Weight and height will be combined to report BMI in kg/m^2
Weist Circunference | Once a year during ten years
  Centimeters in the abdominal circunference

SECONDARY OUTCOMES:
Mental Health and Wellbeing | Once a year during ten years
  Measured with Warwick-Edinburgh Mental Wellbeing Scales questionarie
Coginitive flexibility | Once a year during ten years
  Measured with Impulsive Behavior Scale questionaire

CONTACTS AND LOCATIONS:
Overall Officials: Guillem Jabardo Camprubí, PhD, Principal Investigator — Faculty of Health Science at Manresa

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chooi YC, Ding C, Magkos F. The epidemiology of obesity. Metabolism. 2019 Mar;92:6-10. doi: 10.1016/j.metabol.2018.09.005. Epub 2018 Sep 22. PMID 30253139
- [Background] Baillot A, Vallee CA, Mampuya WM, Dionne IJ, Comeau E, Meziat-Burdin A, Langlois MF. Effects of a Pre-surgery Supervised Exercise Training 1 Year After Bariatric Surgery: a Randomized Controlled Study. Obes Surg. 2018 Apr;28(4):955-962. doi: 10.1007/s11695-017-2943-8. PMID 28963710
- [Background] Lier HO, Biringer E, Stubhaug B, Tangen T. The impact of preoperative counseling on postoperative treatment adherence in bariatric surgery patients: a randomized controlled trial. Patient Educ Couns. 2012 Jun;87(3):336-42. doi: 10.1016/j.pec.2011.09.014. Epub 2011 Oct 27. PMID 22035647